CLINICAL TRIAL: NCT02345824
Title: Early-Phase Study to Assess Tumor Pharmacokinetics and Efficacy of the CDK4/6 Inhibitor Ribociclib (LEE011) in Patients With Recurrent Glioblastoma or Anaplastic Glioma
Brief Title: Early-Phase Study to Assess Inhibitor Ribociclib in Patients With Recurrent Glioblastoma or Anaplastic Glioma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Virginia (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Camilo E. Fadul, MD, Professor, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D13223; 18729 (Other: IRB)
Record Dates: First submitted 2015-01-02; First posted 2015-01-26 (Estimated); Last update posted 2018-06-07 (Actual); Status verified 2018-06

CONDITIONS: Glioblastoma; Glioma
Keywords: CDK4/6 Inhibitor; LEE011; Recurrent Glioblastoma; Anaplastic Glioma; Ribociclib
MeSH Terms: conditions — Glioblastoma; Glioma | interventions — ribociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ribociclib (LEE011) Treatment (Experimental): Patients will be treated with ribociclib (LEE011) (recommended phase 2 dose of 600 mg/day) for 8-21 days prior to surgery. For preliminary evaluation of efficacy and toxicity, patients with Rb-positive tumors will resume treatment with ribociclib at 14-28 days post-surgery on a schedule of 21 days on, 7 days off in a 28-day cycle. Patients will be treated until unacceptable toxicity is observed, or until disease progression as assessed by radiographic or clinical metrics.
  Interventions: Drug: Ribociclib

INTERVENTIONS:
Drug: Ribociclib — CDK4/6 INHIBITOR
  Other Names: LEE011

SUMMARY:
This is a single-institution, open-label, early-phase study to assess the ability of ribociclib (LEE011) to inhibit CDK4/CDK6/Rb/E2F signaling and cell proliferation/viability in core and infiltrating tumor tissues obtained from patients with recurrent glioblastoma or anaplastic glioma compared to the baseline/primary pathologic tumor specimen. Abundant preclinical evidence indicates that Rb-deficient cancer cells are resistant to CDK4/6 inhibition and ongoing trials with CDK4/6 inhibitors exclude patients with Rb-deficient tumors. The investigators will evaluate 10 patients with Rb-positive glioblastoma or anaplastic glioma in this study. Given that a minority of glioblastomas ha Rb loss the investigators anticipate enrolling a maximum of 20 patients, to meet our goal of 10 patients with Rb-positive tumors.

DETAILED DESCRIPTION:
Preliminary evaluation of efficacy and determination of the ribociclib safety profile in patients with brain tumors will be studied. All patients will be treated with ribociclib (600 mg/day) for 8-21 days before surgical resection of the recurrent tumor. Rb status of the recurrent tumor will be determined by immunohistochemistry within 2 weeks after surgery. Patients with Rb-positive tumors will continue treatment with ribociclib (21 days on, 7 days off) after surgery. Patients will be treated until unacceptable toxicity is observed, or until disease progression as assessed by radiographic or clinical metrics. We will determine whether molecular markers associated with changes induced by ribociclib treatment in tumors (matching initial vs. recurrent tumors) correlate with progression-free survival.

Approximately 20% of patients with recurrent high-grade glioma will undergo surgical resection of their tumor typically at the time of first recurrence. These patients will be eligible for this study. An extra 10 mL of blood will be collected during a routine clinical procedure prior to initiation of ribociclib treatment (i.e., baseline blood sample), separated into plasma and buffy coat fractions, and frozen for pharmacokinetic (PK) analysis. Patients will be treated with ribociclib for 8-21 days prior to surgery to identify drug effects on tumor cells, and to determine drug PK. The last presurgical dose of ribociclib will be administered on the day of surgery at 4-8 hours prior to surgery to allow sufficient time for the drug to enter tumor cells, inhibit CDK4/6, and modulate downstream effectors. Blood will be acquired within 1 hour before surgery (as close to the time of surgery as possible). Blood will be separated into plasma and buffy coat fractions, and frozen. During surgery, samples of brain tumor core and infiltrating brain tumor will be acquired. Tissue samples will be frozen or fixed in paraffin embedded blocks and histology for PK and molecular analyses.

ELIGIBILITY:
Inclusion criteria:

* Written informed consent must be obtained prior to any screening procedures
* Patients age 18-85 are eligible for study participation
* History of grade III or IV glioma (GBM or AG) with archived FFPE and/or frozen tumor tissue available
* Patient must be a candidate for surgical resection of recurrent high-grade glioma
* Karnofsky Performance Scale score ≥ 70.
* Life expectancy of 4 months or longer.
* Received at least 1 prior systemic therapy for glioma.
* A sufficient interval must have elapsed between the last dose of prior anti-cancer therapy (including cytotoxic and biological therapies and major surgery) and enrollment, to allow the effects of prior therapy to have abated
* Patients must have adequate organ function
* For continued ribociclib treatment after surgery, immunohistochemical (IHC) confirmation of Rb expression in ≥50% of malignant tumors cells in at least 1 tumor specimen is

Exclusion criteria:

* Impairment of gastro-intestinal (GI) function or GI disease that may significantly alter the absorption of ribociclib such as patients with a history of GI surgery which may result in intestinal blind loops and patients with clinically significant gastroparesis, unresolved nausea, vomiting, or diarrhea of CTCAE grade > 1
* Impaired cardiac function or clinically significant cardiac diseases
* Patients who are currently receiving treatment (within 5 days prior to starting study drug) with agents that are metabolized predominantly through CYP3A4 and that have a narrow therapeutic window. Agents including vitamins, supplements, and herbal supplements that are either (i) metabolized solely through CYP3A4/5, CYP1A2 or BSEP and have a narrow therapeutic window or (ii) are strong inhibitors of CYP3A4/5, CYP1A2 or BSEP. Agents that are known strong inducers or inhibitors CYP3A4 are prohibited. Patients must avoid consumption of grapefruit, Seville oranges or products containing the juice of each during the entire study and for 7 days before the first dose.
* Patients with concurrent severe and/or uncontrolled concurrent medical conditions that the investigator believes could compromise participation in the study (e.g., uncontrolled hypertension and/or diabetes mellitus, clinically significant pulmonary disease, clinically significant neurological disorder, active or uncontrolled infection)
* Pregnant or lactating women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test (> 5 mIU/mL).
* Women of childbearing potential, defined as all women physically capable of becoming pregnant, unless they are using effective methods of contraception during dosing of study treatment. Effective contraception must be used by both sexes (female patients and their male partners) during study treatment and for 30 days after the last dose of study medication
* Fertile males must be willing to use contraception. Fertile males must use condom with spermicide (double barrier method). Effective contraception, as defined above, must be used by both sexes (male patients and their female partners) during study treatment and for 30 days after the last dose of study medication. A condom is required to be used by vasectomized men in order to prevent delivery of the study drug via seminal fluid.
* Patients unwilling or unable to comply with the protocol
* Known diagnosis of human immunodeficiency virus (HIV) or hepatitis C (testing is not mandatory)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2016-03; Primary Completion 2019-09 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Inhibition of CDK4/CDK6 Signaling Pathway in Cell Proliferation | an expected average of 1 year to allow laboratory quality assessment of tumor proliferation
  Levels of phospho-Rb in tumor cells, the fraction of Ki67-positive tumor cells, and the fraction of TUNEL-positive tumor cells in primary (baseline) vs. recurrent (post-LEE011) tumor samples will be assessed via laboratory practices as a means of studying Inhibition of CDK4/CDK6 Signaling Pathway in Cell Proliferation.

SECONDARY OUTCOMES:
Ribociclib Concentration in Tissues | 1 Day Collection as the time of initial surgery
  Concentrations of ribociclib will be gathered from tumor core and infiltrating tumor tissue which is gathered at the time of initial surgery for the removal of the patients tumor.
  This will be completed to assess whether ribociclib treatment induces changes in brain tumor cell fate (proliferation, apoptosis, senescence) and E2F activation. Biomarkers will be compared in ribociclib-treated recurrent tumors vs. matching baseline tumors vs. archived recurrent tumors from other patients.
  Laboratory will assess the frequencies of Rb mutations and loss in primary and recurrent brain tumors.
Ribociclib Concentration in Plasma | time of Pharmacokinetic draws
  Concentrations of ribociclib in blood plasma will be gathered through pharmacokinetic draws at specified time points throughout study participation and will be used to assist in the assessment of whether ribociclib treatment induces changes in brain tumor cell fate (proliferation, apoptosis, senescence) and E2F activation. Biomarkers will be compared in ribociclib-treated recurrent tumors vs. matching baseline tumors vs. archived recurrent tumors from other patients.
  To determine the frequencies of Rb mutations and loss in primary and recurrent brain tumors.
Tumor Progression | Over 1 year, which is expected average length of participation per patient
  Preliminary rates of progression-free survival in patients with high-grade gliomas treated with ribociclib will be measured through radiographic and clinical response metrics, specifically Response Assessment in Neuro-Oncology (RANO) criteria and investigator discretion.
Survival Outcomes | Over 1 year, which is expected average length of participation per patient
  Overall survival in patients with high-grade gliomas treated with ribociclib will be assessed by medical record review and survival follow up.
Ribociclib Safety Profile | 30 days post last dose of LEE011 per patient
  Common Toxicity Criteria Adverse Event (CTCAE 4.0) will be utilized to review ribociclib treatment effects in patients with brain tumors.

OTHER OUTCOMES:
Identifying Treatment Induced Changes in Oncogenic Pathways | Over 1 year, which is expected average length of participation per patient
  To identify treatment-induced changes in compensatory oncogenic pathways that may promote drug resistance, through the use of reverse-phase protein array analysis of tumor samples.
Ribociclib Concentrations in Cerebrospinal Fluid (CSF) | 1 Day Collection as the time of initial surgery
  Cerebrospinal Fluid (CSF) obtained at the time of surgery and processed to assess the amount of ribociclib concentrations

CONTACTS AND LOCATIONS:
Overall Officials: Camilo Fadul, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia Health System, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Miller TW, Traphagen NA, Li J, Lewis LD, Lopes B, Asthagiri A, Loomba J, De Jong J, Schiff D, Patel SH, Purow BW, Fadul CE. Tumor pharmacokinetics and pharmacodynamics of the CDK4/6 inhibitor ribociclib in patients with recurrent glioblastoma. J Neurooncol. 2019 Sep;144(3):563-572. doi: 10.1007/s11060-019-03258-0. Epub 2019 Aug 9. PMID 31399936